CLINICAL TRIAL: NCT02405481
Title: SEPA III: The Effectiveness Trial
Acronym: SEPA III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Nilda Peragallo Montano, Dean and Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20120037
Record Dates: First submitted 2015-03-24; First posted 2015-04-01 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: HIV Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait List Control (No Intervention)
- SEPA III Intervention (Experimental): SEPA brings together two important theoretical perspectives that will be effective and sustainable for HIV/AIDS prevention among Hispanic women in an inner city environment. The content and learning strategies of SEPA are based on the social cognitive theory and of HIV/AIDS prevention that prior research has shown to be the most effective in increasing HIV/AIDS prevention behaviors, modified to take into account the special needs of Hispanic women related to gender inequality and cultural values and practices. SEPA's conceptual framework integrates the Social Cognitive Model of behavioral change with Freire's Pedagogy of the Oppressed that guides the delivery and contextual tailoring.
  Interventions: Behavioral: SEPA III

INTERVENTIONS:
Behavioral: SEPA III
  Arms: SEPA III Intervention

SUMMARY:
The study evaluates the effectiveness of SEPA (Salud, Educacion, Prevencion y Autocuidado; Health, Education, Prevention and Self-Care) to increase HIV prevention behaviors and to reduce the incidence of STIs for Hispanic women when delivered in a real-world setting by community agency personnel. The study recruits Hispanic women between the ages of 18 and 50 who are sexually active and are randomized to either SEPA or a Wait-List Control condition.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic Women,
* 18 to 50 years old,
* Sexually active in the past three months

Exclusion Criteria:

* Non-Hispanic,
* younger than 18,
* older than 50,
* not sexually active

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Condom Use | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nilda Peragallo Montano, DrPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States